CLINICAL TRIAL: NCT06325787
Title: Long-term Comparison of Image-guided Thermal Ablation vs. Lobectomy for Solitary Papillary Thyroid Microcarcinoma: A Multicenter Retrospective Study
Brief Title: Image-guided Thermal Ablation vs. Lobectomy for Solitary Papillary Thyroid Microcarcinoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Yu-kun Luo, Director, Head of Department of Ultrasound, Chinese PLA General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S2021-211-02
Record Dates: First submitted 2024-03-16; First posted 2024-03-22 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Papillary Thyroid Cancer
MeSH Terms: conditions — Thyroid Cancer, Papillary

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- lobectomy (Active Comparator): thyroid lobectomy, is recommended as first-line treatment for papillary thyroid micraocarcinima
  Interventions: Procedure: thyroid lobectomy
- image-guided thermal ablation (Experimental): radiofrequency ablation or microwave ablation
  Interventions: Procedure: image-guided thermal ablation

INTERVENTIONS:
Procedure: thyroid lobectomy — thyroid lobectomy
  Arms: lobectomy
Procedure: image-guided thermal ablation — radiofrequency ablation or microwave ablation or laser ablation
  Arms: image-guided thermal ablation

SUMMARY:
To evaluate the clinical outcomes of image-guided thermal ablation versus thyroid lobectomy for the treatment of papillary thyroid microcarcinoma

ELIGIBILITY:
Inclusion Criteria:

1. solitary papillary thyroid carcinoma confirmed by fine-needle aspiration or core-needle biopsy;
2. largest diameter ≤10 mm;
3. no evidence of extrathyroidal extension( no signs of unsmooth thyroid capsule or involvement of the perithyroidal tissue) on ultrasound;
4. no evidence of cervical lymph node metastasis on US or neck CT;
5. no distant metastasis on chest CT;
6. no history of neck irradiation.

Exclusion Criteria:

* (1)aggressive subtype of papillary thyroid microcarcinoma confirmed by biopsy(1); (2)multiple tumors; (3) incomplete data or lost follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1021 (Actual)
Dates: Start 2013-05-01 (Actual); Primary Completion 2017-01-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
disease progression | more than 5 years
  cervical lymph node metastases, recurrent tumors and persistent tumors
disease-free survival | more than 5 years
  disease-free survival calculated from treatment initiation to disease progression or the last follow-up date

SECONDARY OUTCOMES:
complications | 1 week
  complications after surgery or ablation
procedure time | 1 hour after treatment
  Ablation procedure time was defined from US evaluation for the design of insertion way to treatment terminated. Lobectomy procedure time was defined from incision to closure, not including the anesthesia time.
cost | 1 week
  The ablation cost included preoperative examinations, treatment, local anesthesia and ablation needle costs. The lobectomy cost included preoperative examinations, treatment, general anesthesia, hospital bed, nursing and postoperative medication
estimated blood loss | 1 hour
  estimated blood loss after surgery or ablation
hospitalization | 1 week
  hospitalization for surgery or ablation

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available because of the patients privacy.